CLINICAL TRIAL: NCT05357508
Title: Protocol Title: Colorectal Cancer Screening Decisions Based on Predicted Risk: the PREcision ScreENing Randomized Controlled Trial (PRESENT)
Brief Title: Colorectal Cancer Screening Based on Predicted Risk
Acronym: PRESENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRESENT STUDY
Record Dates: First submitted 2022-04-19; First posted 2022-05-03 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Screening; Personalized Risk; Risk Communication; Shared Decision Making; Screening Behavior
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the Intervention group receive a brochure with their personalized risk score for colorectal cancer and screening recommendations (FIT or colonoscopy) corresponding to their risk level.
  Interventions: Behavioral: Intervention brochure
- Usual care group (Active Comparator): Participants in the Usual care group receive the standard brochure designed by the Vaud screening program. This brochure recommends screening to all individuals beginning at age 50 and presents both FIT and colonoscopy as equal options.
  Interventions: Behavioral: Control brochure

INTERVENTIONS:
Behavioral: Intervention brochure — Provide participants with information about their personalized risk for colorectal cancer and appropriate screening recommendations to facilitate their screening option choice.
  Arms: Intervention group
Behavioral: Control brochure — Provide participants with general information about options for colorectal cancer screening.
  Arms: Usual care group

SUMMARY:
The primary objective is to study the effect of communicating individual CRC risk score and screening recommendations on appropriate screening uptake at six months in individuals at low, moderate and high risk of developing CRC.

The secondary objectives:

* Assess the feasibility of a subsequent larger RCT designed to detect a change in clinical outcomes;
* Explore the impact of psychological factors (perceived susceptibility for CRC, perceived benefits from and barriers to screening) on appropriate screening uptake and participation rates.

The investigators will perform a pilot randomized controlled trial (RCT) of 880 residents from the canton Vaud (Switzerland) aged between 50 and 69 years. The QCancer calculator will be used to calculate the personalized risk score. The participants in the intervention group will receive a brochure with a personalized risk score and appropriate screening recommendations. The participants in the control group will receive the standard brochure of the Vaud CRC screening program, regardless of participants' risk level. Six months after the intervention, the investigators will measure the proportion of the participants who have undergone appropriate screening. Screening will be considered as appropriate if participants at high risk undertake colonoscopy and participants at low risk undertake FIT. Both tests are appropriate for participants at moderate-risk. The hypothesis is that in the intervention group, individuals will be more likely to undergo screening appropriate to a participant's individual risk level, whereas the choice of the screening test in the control group will not differ between risk levels.

This study should advance the field of risk-based screening. This may give insights about how to optimize CRC screening programs and offer to the population screening options with a better risk-benefit balance.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) can be effectively prevented by screening. Risk to develop CRC within 15 years is related to increasing age, sex, family history, and lifestyle and, thus, can vary from <1% to >15%.

Fecal immunochemical test (FIT) and colonoscopy are the most widely used screening tests. Colonoscopy is the most accurate test, but is related to risks of bleeding and perforation. Colonoscopy resources are limited, and high uptake of screening colonoscopy for low-risk individuals can cause long wait times for those with CRC symptoms or positive FIT. FIT is less costly can be done at home without preparation and, if done regularly, prevents most CRC mortality, especially in moderate and low-risk individuals. To offer the screening options with a reasonable risk-benefit balance, FIT should be recommended to individuals at low (<3% to develop CRC in 15 years) and moderate (3-6%) risk, and colonoscopy to those at high (>6%) risk.

The primary objective is to study the effect of communicating individual CRC risk score and screening recommendations on appropriate screening uptake at six months in individuals at low, moderate and high risk of developing CRC.

The secondary objectives:

* Assess the feasibility of a subsequent larger RCT designed to detect a change in clinical outcomes;
* Explore the impact of psychological factors (perceived susceptibility for CRC, perceived benefits from and barriers to screening) on appropriate screening uptake and participation rates.

The investigators will perform a pilot randomized controlled trial (RCT) of 880 residents from the canton Vaud (Switzerland) aged between 50 and 69 years. The QCancer calculator will be used to calculate the personalized risk score. The participants in the intervention group will receive a brochure with a personalized risk score and appropriate screening recommendations. The participants in the control group will receive the standard brochure of the Vaud CRC screening program, regardless of the participant's risk level. Six months after the intervention, the investigators will measure the proportion of the participants who have undergone appropriate screening. Screening will be considered as appropriate if participants at high risk undertake colonoscopy and participants at low risk undertake FIT. Both tests are appropriate for participants at moderate-risk. The hypothesis is that in the intervention group, individuals will be more likely to undergo screening appropriate to participant's individual risk level, whereas the choice of the screening test in the control group will not differ between risk levels.

This study should advance the field of risk-based screening. This may give insights about how to optimize CRC screening programs and offer to the population screening options with a better risk-benefit balance.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 and 69;
* Residents of the Canton of Vaud;
* Have signed an informed consent (paper or electronic).

Exclusion Criteria:

* Current CRC symptoms;
* Personal CRC history;
* In colonoscopy surveillance for follow-up of high-risk polyp(s);
* Inflammatory bowel disease;
* Having done a colonoscopy within 9 years or a FIT within 1,5 years;
* Planning to leave Switzerland definitively within the next six months.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Self-reported appropriate screening uptake | 6-8 months after the intervention
  Proportion who completed screening test appropriate to risk level. For low risk (<3% 15-yr CRC risk), completing a FIT. For intermediate risk (3-6%15-yr CRC risk), completing a FIT, completing a colonoscopy, or having a colonoscopy appointment. For high risk (>6% 15-yr CRC risk), completing a colonoscopy or having a colonoscopy appointment.

SECONDARY OUTCOMES:
Self-reported overall screening participation | 6-8 months after the intervention
  Proportion who completed any CRC screening test (FIT, colonoscopy, colonoscopy appointment, CT colonography, blood test, etc.
Participation in the randomized trial | 6 weeks after mailed invitations
  Proportion of those invited with completed paper or electronic consent
Eligibility for the Vaud CRC screening program | 6 weeks after mailed invitations
  Proportion of those who returned the baseline questionnaire who are eligible for the Vaud screening program (i.e. not up-to-date with screening, not in colonoscopy surveillance, no personal CRC history, etc.)
Self-reported anxiety | 6 weeks after mailed invitations
  Mean anxiety score using adapted questions from a standardized questionnaire (STAI Fr)
Linkage to Vaud CRC screening program | 3-6 months after measurement of primary outcome
  Proportion of study participants who consent and whose screening status are obtained from the Vaud CRC screening program
Linkage to Vaud tumor registry | 6 months to 10 years after measurement of primary outcome
  Proportion of study participants who consent and whose cancer status are obtained from the Vaud tumor registry. Long time frame chosen given considerable delay in updating the tumor registry and interest in cancer outcomes several years after measurement of primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Selby, MD, MAS, Principal Investigator — Center for Primary Care and Public Health (Unisanté)
Locations (1):
- Center for Primary Care and Public Health (Unisante), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of the primary results, the data that support the findings of this study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Will become available upon publication of the primary results and remain available 5 years.
Access Criteria: Reasonable request to the principal investigator

REFERENCES:
- [Background] Hippisley-Cox J, Coupland C. Development and validation of risk prediction algorithms to estimate future risk of common cancers in men and women: prospective cohort study. BMJ Open. 2015 Mar 17;5(3):e007825. doi: 10.1136/bmjopen-2015-007825. PMID 25783428
- [Background] Samusure J, Horisberger D, Diserens C, Ducros C, Auer R, Bodenmann P, Durand MA, Selby K. [Information materials for colorectal cancer screening for citizens with low health literacy]. Rev Med Suisse. 2022 Mar 30;18(775):616-620. doi: 10.53738/REVMED.2022.18.775.616. French. PMID 35353458
- [Background] Plys E, Bulliard JL, Chaouch A, Durand MA, van Duuren LA, Brandle K, Auer R, Froehlich F, Lansdorp-Vogelaar I, Corley DA, Selby K. Colorectal Cancer Screening Decision Based on Predicted Risk: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 7;12:e46865. doi: 10.2196/46865. PMID 37676720
- [Derived] Plys E, Bulliard JL, Chaouch A, Durand MA, van Duuren LA, Braendle K, Auer R, Froehlich F, Lansdorp-Vogelaar I, Corley DA, Selby K. Colorectal Cancer Screening Based on Predicted Risk: A Randomized Controlled Trial. Am J Gastroenterol. 2025 Oct 1;120(10):2432-2439. doi: 10.14309/ajg.0000000000003311. Epub 2025 Jan 7. PMID 39774118
- See also: Risk calculator used — https://qcancer.org/15yr/colorectal/index.php